CLINICAL TRIAL: NCT00869193
Title: Effect of Grape Seed Extract High in Polyphenols on Blood Pressure in Subjects With Elevated Blood Pressure Levels
Brief Title: Effect of Grape Seed Extract on Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Collaborators: University of Edinburgh (Other)
Responsible Party: Rouyanne Ras, Unilever R&D Vlaardingen
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 08050V
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Last update posted 2009-08-28 (Estimated); Status verified 2009-08

CONDITIONS: Elevated Blood Pressure
Keywords: Blood pressure; Grape seed
MeSH Terms: conditions — Hypertension | interventions — Grape Seed Extract; Polyphenols; microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Grape seed (Active Comparator): Grape seed extract
  Interventions: Dietary Supplement: Grape seed extract
- Placebo (Placebo Comparator): Microcrystalline cellulose
  Interventions: Dietary Supplement: Microcrystalline cellulose (placebo)

INTERVENTIONS:
Dietary Supplement: Grape seed extract — Subjects will daily consume one capsule with grape seed extract for 8 weeks.
  Other Names: Polyphenol
  Arms: Grape seed
Dietary Supplement: Microcrystalline cellulose (placebo) — Subjects will daily consume one capsule with microcrystalline cellulose for 8 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether an 8-week intervention with grape seed extract is effective in reducing daytime ambulatory blood pressure in male and postmenopausal female with elevated daytime blood pressure values.

DETAILED DESCRIPTION:
Background: High blood pressure is a major risk factor for morbidity and mortality from stroke, heart disease, and end-stage renal disease. Several studies have shown that dietary polyphenols derived from fruits and vegetables (including those from grape products) can lower blood pressure in both normotensive and hypertensive subjects.

Study objectives: Primary objective: To study, in subjects with elevated blood pressure levels, the effects of grape seed extract high in polyphenols, on daytime ambulatory systolic and diastolic blood pressure (SBP and DBP, respectively). Secondary objective: To explore mechanistic pathways responsible for the blood pressure lowering efficacy in case a blood pressure lowering effect is shown.

Study population: Each treatment group will consist of 35 men and postmenopausal women (35-75 years of age) with daytime SBP between 120 and 159 mmHg. The total number of subjects will be 70.

Study design: This study will have a randomized, double-blind, placebo-controlled parallel design with 2 treatments, a 1-week run-in period, and an 8-week intervention period. The 2 treatments will consist of placebo capsules and capsules with grape seed extract.

Study outcomes: Daytime ambulatory blood pressure (ABP) will be measured every 20 minutes for 2 x 12 hours at baseline and 2 x 12 hours at the end of intervention. Furthermore, before and after the intervention period, 24-hour urine will be collected and 2 blood samples will be taken in order to investigate mechanistic pathways and platelet function.

ELIGIBILITY:
Inclusion Criteria:

* Male and postmenopausal female subjects in the age ≥ 35 and ≤ 75 at start of the study
* BMI ≥ 18.5 and ≤ 30.0 kg/m2
* Apparently healthy: no reported diseases that may affect study results and pre-selected blood parameters within normal range
* Informed consent signed
* Willing to refrain from supplements, food products, diets and drugs that may interfere with the outcomes of the study

Exclusion Criteria:

* Mean of 6-hour ambulatory SBP < 120 mmHg, > 159 mmHg and/or DBP > 99 mmHg
* 10-year risk mortality risk on CVD > 10% according to NHG standard M84. For subjects > 65 years of age and SBP ≥ 140 mmHg the study physician will assess eligibility
* Irregular pulse or pulse < 50 or > 100 bpm
* Intense exercise >10 h/w
* Reported weight loss/gain > 10% of body weight in the 6 month preceding pre-study examination
* The habit of smoking during the past year

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Difference between treatment and placebo in changes from baseline of ambulatory systolic and diastolic blood pressure | 8 weeks of intervention

SECONDARY OUTCOMES:
Difference between treatment and placebo in changes from baseline of mechanistic markers in plasma and/or urine (vasoactive factors and markers of polyphenol metabolism) and platelet function (only measured in case of a relevant BP-lowering effect) | 8 weeks of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Rouyanne T Ras, Msc, Principal Investigator — Unilever R&D Vlaardingen
Locations (1):
- Unilever R&D Vlaardingen, Vlaardingen, Netherlands